CLINICAL TRIAL: NCT02552459
Title: Effect of Dexmedetomidine Combined With Sufentanil for Postoperative Intravenous Analgesia in Neurosurgery: A Randomized Controlled Study
Brief Title: Effect of Dexmedetomidine Combined With Sufentanil for Postoperative Intravenous Analgesia in Neurosurgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xinxin Shao, resident, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FirstSunYetSen-jn2015
Record Dates: First submitted 2015-05-26; First posted 2015-09-17 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Arteriovenous Malformation
Keywords: dexmedetomidine; patient controlled analgesia
MeSH Terms: conditions — Arteriovenous Malformations | interventions — Sufentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- sufentanil (Active Comparator): sufentanil 150μg，intravenous administration during the following 72 hours after operation.
  Interventions: Drug: Sufentanil
- sufentanil&dexmedetomidine 1 (Experimental): sufentanil 150μg，dexmedetomidine 0.05μg/kg/h，intravenous administration during the following 72 hours after operation.
  Interventions: Drug: Sufentanil; Drug: dexmedetomidine 1
- sufentani&dexmedetomidine 2 (Experimental): sufentanil 150μg，dexmedetomidine 0.1μg/kg/h，intravenous administration during the following 72 hours after operation.
  Interventions: Drug: Sufentanil; Drug: dexmedetomidine 2
- sufentanil&dexmedetomidine 3 (Experimental): sufentanil 150μg，dexmedetomidine 0.15μg/kg/h ，intravenous administration during the following 72 hours after operation.
  Interventions: Drug: Sufentanil; Drug: dexmedetomidine 3

INTERVENTIONS:
Drug: Sufentanil — sufentanil 150μg， intravenous administration during post-operative 72 hours.
  Other Names: Sufentanyl
Drug: dexmedetomidine 1 — dexmedetomidine 0.05μg/kg/h, Continuous intravenous injection for 72 hours after operation
  Other Names: Dex,Dexmedetomidine
  Arms: sufentanil&dexmedetomidine 1
Drug: dexmedetomidine 2 — dexmedetomidine 0.1μg/kg/h, Continuous intravenous injection for 72 hours after operation
  Other Names: Dex,Dexmedetomidine
  Arms: sufentani&dexmedetomidine 2
Drug: dexmedetomidine 3 — dexmedetomidine 0.15μg/kg/h, Continuous intravenous injection for 72 hours after operation recorded in the following 72h.
  Other Names: Dex,Dexmedetomidine
  Arms: sufentanil&dexmedetomidine 3

SUMMARY:
The purpose of this study is to determine effect of combined medication of sufentanil and dexmedetomidine in patient controlled analgesia after neurosurgery.

DETAILED DESCRIPTION:
Sufentanil is a classical drug for postoperative analgesia. Dexmedetomidine is a commonly used α2-adrenergic receptor, and it helps provide sedation, analgesia and inhibition of sympathetic activation. The investigators propose to recruit 120 patients who is undergoing the arteriovenous malformation embolism operation in department of Neurosurgery. Patients will be randomly divided into 4 groups(control group, sufentanil and low dexmedetomidine dose group, sufentanil and middle dexmedetomidine dose group, sufentanil and high dexmedetomidine dose group), then the investigators select post-operative records to determine whether dexmedetomidine can take a positive role in neurosurgical analgesia.

ELIGIBILITY:
Inclusion Criteria:

1. patients undergoing venous malformation embolization operation through general anesthesia.
2. aged 18-65 years old.
3. operating time varies 1-4h,and extubation after the operation.

Exclusion Criteria:

1. long-term use of analgesics,sedatives or non steroidal anti-inflammatory drugs history.
2. known for dexmedetomidine or other drugs allergy in this study.
3. cannot communicate.
4. preoperative systolic blood pressure <90 mmHg, or the heart rate <50/min.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pain on the VAS scale | within the following 72 hours after surgery
  measure the VAS score at pre-operative day and post-operative 4h、8h、12h、24h、48h、72h。

SECONDARY OUTCOMES:
blood pressure(BP)(mmHg) | within the following 72 hours after surgery
  measure BP(mmHg),HR (/min),spO2(%), and breath(/min),on pre-operative day and at post-operative 4h、8h、12h、24h、48h、72h
heart rate(HR) (/min) | within the following 72 hours after surgery
  measure BP(mmHg),HR (/min),spO2(%), and breath(/min),on pre-operative day and at post-operative 4h、8h、12h、24h、48h、72h
spO2(%) | within the following 72 hours after surgery
  measure BP(mmHg),HR (/min),spO2(%), and breath(/min),on pre-operative day and at post-operative 4h、8h、12h、24h、48h、72h
breath(/min) | within the following 72 hours after surgery
  measure BP(mmHg),HR (/min),spO2(%), and breath(/min),on pre-operative day and at post-operative 4h、8h、12h、24h、48h、72h
sedation level on ramsay sedation score | within the following 72 hours after surgery
  measure sedation level using ramsay sedation score on pre-operative day and at post-operative 4h、8h、12h、24h、48h、72h
vomit times | within the following 72 hours after surgery
  measure vomit times on pre-operative day and at measure sedation level using ramsay sedation score on pre-operative day and at post-operative 4h、8h、12h、24h、48h、72h
nausea | within the following 72 hours after surgery
  measure whether nausea exists on pre-operative day and at measure sedation level using ramsay sedation score on pre-operative day and at post-operative 4h、8h、12h、24h、48h、72h

OTHER OUTCOMES:
dose of rescue tramadol | within the following 72 hours after surgery
  measure the dose of tramadol using as rescue drug on post-operative 24h、48h、72h

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Nan, doctor, Principal Investigator — The First Affiliated Hospital, Sun Yat-sen Unniversity; Shao Xinxin, master, Principal Investigator — The First Affiliated Hospital, Sun Yat-sen Unniversity
Locations (1):
- the First Affiliated Hospital of Sun Yetsen University, Guangzhou, Guangdong, China